CLINICAL TRIAL: NCT07112508
Title: PRISM: The PRimary Care Individual Social Norms MSK Data Dashboard: a Cluster Randomised Feasibility Trial in Clinician Management of Musculoskeletal Patients.
Brief Title: PRISM: The PRimary Care Individual Social Norms MSK Data Dashboard: a Feasibility Trial
Acronym: PRISM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Homerton University Hospital NHS Foundation Trust (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRISM1
Record Dates: First submitted 2025-07-18; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Musculoskeletal Disorders
Keywords: Musculoskeletal; Primary Care; First Contact Physiotherapy; First Contact Practitioner; Digital Health; Behaviour change
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: This is a pragmatic feasibility cluster randomised controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRISM Intervention Group (Experimental): This group will receive the PRISM dashboard on a monthly basis to be discussed in clinical supervision. It will show them where their clinical behaviours sits relative to their patients. The control will be treatment as usual.
  Interventions: Behavioral: PRISM dashboard is a data report
- usual care group (Active Comparator): This group will receive usual care and the clinicians will receive no information about their performance.
  Interventions: Other: THe usual care intervention is a first contact physiotherapy service.

INTERVENTIONS:
Behavioral: PRISM dashboard is a data report — The PRISM dashboard captures a clinicians activity relative to their peers. It provides social norms feedback on an array of clinical interventions that an FCP makes.
  Arms: PRISM Intervention Group
Other: THe usual care intervention is a first contact physiotherapy service. — usual care
  Arms: usual care group

SUMMARY:
Background:

20 million people in UK have musculoskeletal (MSK) aches and pains. They commonly see their GP about this problem, but practices are so busy that it can mean a long wait for appointments. First Contact Practitioner (FCPs) are now working in the GP practices to see patients with MSK problems instead of their GP. A national evaluation has found this to be working well.

For FCPs working in GP practices there is more clinical risk. The patients have not been previously screened by a doctor to ensure there is no medical cause for their pain. The Chartered Society of Physiotherapists (CSP) has advised that all FCPs be clinicians with the highest level of experience, known as Advanced Practitioners. However the demand for FCPs far outweighs the number of Advanced Practitioners available so physiotherapists being hired have less experience.

Evidence shows that clinicians of different experience levels have different decision-making strategies which may cause unwarranted variation in care. A new method is needed for oversight and support of the FCPs. Clinical supervision is commonly utilised in the NHS and in physiotherapy teams. It is a space to reflect on a clinician's performance and create learning opportunities.

This research suggests an individual data dashboard, shared only with individuals and their supervisor, that feeds back a clinician's own decision-making data to them, relative to their peers. For example, the participant is "in the top 20% of MRI requesters" or "in the top 20% of those referring to social prescribing". This type of feedback is known as 'social norms' feedback. It has been proven to be an effective way to change healthcare workers behaviour. The intervention will be called PRISM: Primary Care Individual Social Norms MSK Data Dashboard.

Aims To explore the feasibility of a randomised clinical trial comparing the clinical decision-making behaviour of FCP services using the PRISM Dashboard and a usual service with no clinician feedback.

Design & Methods:

This research is a feasibility trial, a process to assess whether a future full scale clinical trial within the NHS would work. It will take place across 4 different Primary Care commissioning areas to determine the possibility of recruitment, retention, outcome collection and whether people will use the intervention.

PPIE for this research included one primary care PPI rep, one digital interventions PPI rep and 3 Healthwatch PPI reps. Engaging different PPI sources enabled participation from different social , cultural and ethnic backgrounds.

Dissemination I will communicate research updates and outputs in conferences, via social media, blogs, newsletters and podcasts. I will use my own network as well as the reach of collaborators in this work, ie. Healthwatch, NHS England/Improvement, The (CSP), the physiotherapy digital network, Keele University and UCL research networks.

DETAILED DESCRIPTION:
SUMMARY BACKGROUND AND RATIONALE

Over 20 million people in the UK live with a musculoskeletal (MSK) condition; accounting and one in three GP consultations . The Fuller Stocktake Report from NHS England described services as "stretched beyond capacity" with "signs of genuine and growing discontent" . The NHS, in keeping with the international trend to include non GP clinicians in the Primary Care workforce) have incorporated pharmacists, physiotherapists, practice nurses and physician associates within the primary care workforce to address the challenges of capacity and demand.

In the UK, patients with MSK problems consult a First Contact Practitioner (FCP) based in primary care instead of their GP, improving patient access to MSK management and freeing GP capacity . FCPs service in the UK, Sweden and Canada were found to be acceptable and effective in national evaluations .

The Chartered Society of Physiotherapy (CSP) and Health Education England (HEE) called for FCPs to be 'Advanced Practitioners' , a certification conferred officially on those with particular expertise. This was deemed necessary to meet the level of risk associated with having a clinical case load of patients who have not been screened by a doctor. However the pool of APs is limited and less experienced FCPs have been recruited into these posts.

FCPs in GP practices, work alone and lack the peer support of a typical physiotherapy department. Unfortunately, data suggests that less experienced FCPs are less likely to provide evidence-based MSK care. Clinical audits of FCP decision-making in over 2000 patients, from the Midlands and London, shows distinct differences in decision-making where Band 7 FCPs were almost twice as likely as Band 8 colleagues to send the patient to the GP for a second opinion, they underutilised 'social prescribing' and 'shared decision-making tools' and ordered more MRIs than their more experienced colleagues. The appropriate use of skills such as imaging requests and onward referrals should be utilised with consistency and in step with evidence-based guidance.

Evidence suggests supervision, social norms and feedback in clinical contexts can improve care. Specifically, that clinical supervision is an effective aspect of professional training and development that can improve evidence-based practice . It has been shown to support the effectiveness of care and reduce burnout and stress. A Cochrane review highlighted the importance of individual tailored feedback in supervision for learning and improving clinical standards. There have been calls for better use of data related to clinician performance, in clinical supervision eg, data on patient outcomes and experience and service level that show number of patients seen, follow up rates, resource use etc. This data has the potential to improve effectiveness by providing more formal and structured feedback on decision-making and quality of care . Presenting feedback about an individual's position in relation to their peers, ('social norms' feedback) can be used to identify outliers in clinical decision-making and nudge behaviour change. A recent systematic review and meta-analysis showed that social norms interventions are effective in "changing health care practitioner behaviours and improving patient outcomes". They nudge clinician behaviour towards desired standards and reduce variation in care . The potential of social norms interventions remains unexplored in MSK services in Primary Care.

In partnership with the Chartered Society of Physiotherapists and a network of improvement focused FCP services across the country, the investigators have worked to create a dataset that is comprised of retrospective FCP data that the investigators can analyse . Some of this data will be uniform as it was collected through a template in Emis and System one. The data collection template was developed as a collaboration between Keele University, the CSP and NHS digital physiotherapy leaders . Other services collected data through their own digital forms and local methods. They contain primarily the same metrics but with local variation. For the PRISM study the investigators will utilise the template where possible but the investigators can accommodate data that has been collected through multiple methods. As long as the datapoints capture the activity in FCP service, then it can be utilised for individual social norms feedback to FCPs in the PRISM study. This data is routinely available as it is collected for service level analysis. Although service level data enables knowledge at a provider level, it does not address variation in clinician performance or provide a mechanism for individual clinicians to reflect on their decision-making and change behaviour. The PRISM studies have formed a collaboration with industry partner www.VUIT.online.com to develop an interactive data dashboard which the investigators make available to all NHS FCP services.

Research Question:

To assess the feasibility of recruiting and retaining patients and clinicians to the study, collecting patient rated outcome measures and patient rated experience measures and assess the usage of the intervention, so that the investigators determine the feasibility of evaluating the clinical effectiveness and cost effectiveness of the PRISM dashboard in a future clinical trial?

Objectives: 1. To assess the feasibility of recruiting and retaining individuals and FCP teams to the trial.

2. To assess the feasibility of collecting patient rated outcome measures (PROMs) and patient rated experience measures (PREMS)from FCP patients 3. To assess implementation of the data collection template in both arms of the study.

4. To assess engagement of first contact physiotherapists with the PRISM dashboard.

5. To assess the feasibility of measuring effectiveness of clinical supervision from the suprevisees perspective 6. To inform the protocol for a fully powered RCT to determine the clinical and cost-effectiveness of using the PRISM Dashboard and Guidance Document

Type of trial: Phase- Feasibility, single-blind, cluster randomised, parallel group, multi-site trial in Musculoskeletal patients.

FCPs and their supervisors in the intervention group will receive the password protected dashboard monthly via email link. The dashboard will contain visualisations of their clinical decision-making compared with social norms. The dashboard can filter to compare areas with similar index of deprivation.

Participants (FCPs and supervisors) will be given a Guidance Document based on the outputs of WP2. It will contain sections on how to interpret the data, information on evidence-based standards and resources to meet learning needs.

The FCP and their supervisor will review the dashboard in clinical supervision. The data can inform knowledge of the complexity of the caseload, outlier occurrences, common clinical behaviours such as decisions around investigations and referrals onward, as well as the clinicians use of the available spectrum of local services and interventions.

Trial duration per participant: Patient participants : Patient (Baseline, 3FU, 6FU) Clinical participants: Patient (Baseline, 3FU, 6FU)

Estimated total trial duration January 2026-September 30th 2026 Planned trial sites: multi-site. 4 sites Total number of participants planned: Investigators will recruit from 4 clusters with approximately 12 physios per site. Primary care areas will be allocated on a 1:1 basis. The sample of 4 clusters have been selected for the feasibility study as these are the numbers that are feasible to work with within the timelines and capacity of the ACAF award. A samples size calculation for the main trial has not been done as this is beyond the remit of this study.

Statistical methodology and analysis: The trial will be reported in line with CONSORT guidance. Analysis will be done by intention to treat principles based on clusters. Binary and other categorical measures will be summarised using frequencies and percentages. Continuous measures will be summarised using means and standard deviations (or medians and IQRs). All outcome measures will be summarised separately by study arm. Differences in outcomes between arms will be modelled using mixed effects linear or logistic regression models. Potential therapist effect will be assessed using the intraclass correlation coefficient. The precision of estimates will be assessed using 95% confidence intervals

Improvement to current practice It is essential to clearly identify opportunities to ensure that all FCPs can safely work toward MSK best practice standards. The unwarranted variation in care associated with skill deficits and low levels of peer support in the FCP workforce can lead to clinical risk and a negative impact on care. This protocol proposes a Primary Care Individual Social Norms MSK Data Dashboard - PRISM. The dashboard is shared with individual FCPs and their clinical supervisors. It is a social norms behaviour change intervention that aims to nudge clinician behaviour toward evidence-based standards and social norms by telling them, for example, the participant is in "the top 20% of MRI requesters", or "the top 20% of those utilising shared decision-making tools". It will report on the NHS England, 'Quality Safety and Effectiveness' measures for MSK Primary Care. In this case, social norms refers to the appropriate and expected behaviour of FCPs based on the behaviour of the majority and professional standards. This PRISM dashboard will be reviewed as part of supportive clinical supervision., allowing the FCP and their supervisor to discuss the data, reflecting on contextual factors such as caseload complexity, deviations from social norms and potential learning opportunities. By enabling FCPs and clinical supervisors to discover and address the learning needs of a clinical workforce, the investigators are creating a mechanism to identify and address unwarranted variation and thereby improve patient care.

Study design and setting:

This is a pragmatic feasibility cluster randomised controlled trial with embedded qualitative work package (described in WP2).

Setting: the trial will be set in UK general practices who have an FCP service. There is an ideal opportunity to evaluate the PRISM intervention within this existing national network. The study will be listed on the CRN portfolio. City & Hackney Place Based Partnership, Primary Integrated Community Service Nottingham and Sandwell and West Birmingham Hospitals NHS Trust have expressed interest in the PRISM dashboard. Participating FCPs and supervisors will be blinded to their intervention for the first 2 months. After 2 months FCPs in the intervention arm will receive the dashboard and the control arm will not. Patients will be blind as to which group they are in. Outcomes will be collected at Baseline, 3 and 6 months.

Design This is a pragmatic feasibility cluster randomised controlled.

The Intervention The intervention is described in line with the TiDieR template for intervention description(54).

There are four parts to the intervention.

There are four parts to the intervention.

1. Data collection FCP clinical assessment and management data will be collected from FCP Clinics in EMIS and SystemOne for the purpose of comparing an individual clinician's behaviour with the FCP clinician group as a whole. In some cases this data is collected routinely already for service level data analysis. Some clinics use a template that was developed by the Keele MIDAS team with collaboration from the Chartered Society of Physiotherapists and NHS collaborators. This may be in intervention or the control arm. The template is used by FCPs at the end of each consultation and takes a maximum of one minute to complete. It is a summary of the consultation, with each tick-box being linked to the relevant Snomed codes to enable clean data extraction from the consultation record. The same data points can be extracted from services not using the templateThis will involve the same Snomed codes.
2. The PRISM dashboard The PRISM Dashboard will be developed at Keele University with commercial partners VUIT Online. After an initial 8 weeks of data collection, FCPs and their supervisors in the intervention group will receive the password protected dashboard monthly via email link.. The dashboard will feature visual representations of their clinical decision-making, benchmarked against the aggregated data of all FCPs which is presented as the 'social norm'. In behavior change theory, social norms refer to the unwritten rules and expectations about how individuals should behave in specific situations. These norms are shaped by the collective perceptions and behaviors of a group, influencing what is considered appropriate and expected . The dashboard can filter to compare areas with similar index of deprivation, unemployment etc. The dashboard will compare behaviours relative to the full scope of available interventions, creating a nudge mechanism for broader use of interventions.
3. The guidebook Participants will be given a Guidance Document based on the outputs of WP2. It will contain sections on how to interpret the data, information on evidence-based standards and resources to meet learning needs. The FCP and their supervisor will review the dashboard in clinical supervision.
4. Structured clinical supervision

The FCP and their supervisor will review the dashboard in clinical supervision. The data will inform knowledge of the complexity of the caseload, outlier occurrences, common challenges such as decisions around imaging or investigations and referrals onwards.

Control: Clinicians in the control group will continue treatment as usual over the trial period but will have no feedback until the trial is over

Recruitment

Sites who express and interest will be given the PIS and assessed in terms of eligibility. If they consent and are eligible, they will be assessed in terms of the feasibility of providing data to the study on a monthly basis. They must have the ability to provide a monthly data upload from the clinical workflow. Data sharing agreements will be in place and the research team will perform an audit of data collection processes. FCPs must be in monthly clinical supervision. Inclusion and Exclusion criteria will be determined by IN, JH and ED

Patient participants: Clinical staff from the CRN will undertake monthly searches of the primary care medical records to identify patients who saw an FCP and upload this data to the UCL ARC Trusted Research environment. Patients will be sent an invitation text followed by a reminder text (or invitation letter if they do not have a mobile number), which contains a link to the participant information leaflet, data privacy statement, consent forms, and online survey. All patients will receive treatment as usual. Inclusion and Exclusion criteria will be determined by IN, JH and ED

PRISM will be a CRN portfolio study. Primary care FCPs teams will be invited to take part via email. Screening will be completed by the CI. Participant sites will be recruited through the FCP network.

Participant recruitment at a site will only commence when the trial has

1. Been initiated by the Sponsor (or its delegated representative), and
2. Issued with the 'Open to Recruitment' letter or Green Light letter from the Sponsor.

A screening log will be kept and maintained to monitor recruitment.

Consent Site consent will be obtained from the FCP service lead. The FCP service lead will be given the Information Sheet and provided with an opportunity to ask questions. 2 weeks will be given for consideration by the site before taking part. The two-week period reflects the fact that multiple persons may need to be consulted before a decision to consent is made. It will be recorded in the trial record when the Information sheet is given. Site consent will ultimately be taken by the CI. If consent is not given, the site will be invited to give feedback as to why but this is not required. Any feedback will be recorded as part of the CONSORT process.

Individual consent will be obtained by a GCP accredited researcher, either the CI, research assistant or a suitably qualified and experienced person. For individual consent a week for consideration will be given. The participant will have the opportunity to ask questions. It will be recorded in the medical/case notes/source documents when the participant information sheet (PIS) has been given to the participant. The Investigator will explain that participants are under no obligation to enter the trial and that they can withdraw at any time during the trial, without having to give a reason.

No clinical trial procedures will be conducted prior to the participant giving consent by signing the consent form. Consent will not denote enrolment into trial.

A copy of the signed informed consent form will be given to the participant. The original signed form will be retained in the trial file at site and a copy placed in the medical/case notes/source documents.

The PIS and consent form will be reviewed and updated if necessary throughout the trial (E.g: where new safety information becomes available) and participants will be re-consented as appropriate.

TRIAL PROCEDURES

Sites

* Sites will be assessed for eligibility
* Site consent will be taken
* Consent from participating clinicians will be taken
* The data extraction will be conducted by the NHS team who are the data custodians of the data. They will be responsible for fully anonymising the data The personal identified data will be deleted, including a process of changing postcode to IMD and DOB to age. The clinician identifier will remain in the data
* Data collection from each site will be monthly and a secure link to the UCL ARC Trusted Research Environment will facilitate this.
* The intervention will be provided on a monthly basis to clinicians
* Clinical supervision will also be held on a monthly basis

Patient participants will all receive only treatment as usual.

1. After an FCP appointment is booked the investigators will use the CRN to identify who has been booked for an FCP appointment and 20% of patients will be contacted.
2. If a patient is eligible and consents to participate, outcome measures will be digitally sent to them for completion or taken by the Research Assistant on this study by phone if the patient prefers.
3. Baseline visit will occur within 14 days of the FCP appointment.
4. Follow up will be scheduled for 3 months and 6 months

If patient outcomes fall outside the preferred time window, the investigators collect them anyway as there may be important feasibility learning re outcomes.

Randomisation

Clusters will be randomised to the intervention or control by a statistician independent to the study, including stratification based on compiled general practice list size to allocate in a ratio of 1:1 (2 intervention, 2 control). A statistician will computer-generate the random sequence and ensure concealment by providing each place an anonymised code. Allocation will be shared with the study team.

It was decided to randomise by Primary Care locality rather than by practice or primary care network as the risk of intervention contamination between the intervention and control group was too great if they were within the same clinical teams.

Randomisation will be provided by a PRIMENT statistician who is blinded to the trial. It will be set up, tested and validated following Priment SOPs.

Schedule of events

The schedule of procedures for the Site team is as follows

* Initial visit to launch site.
* Collect and anonymise the FCP data monthly and submit to UCL ARC Trusted Research Environment
* Visit to support site in first 8 weeks
* Assessment of outcome measure collection
* Assessment of any local risks

Data Management

A data management plan will be created which will include details of the data collection tools, methods of completing case report forms, sign off of completed CRFs, source document identification and methods to maximise completeness of data collection.

It will be the responsibility of the investigator to ensure the accuracy of all data entered in the CRFs. The delegation log will identify all those personnel with responsibilities for data collection and handling, including those who have access to the trial database.

Data collected for the study will be entered in the medical/case notes/source documents in the first instance and then transcribed into the CRFs.

All data will be collected and handled in accordance with Priment SOP Data Handling and the trial specific arrangements will be detailed in the data management plan.

The CRFs will be entered into a web-based clinical data management system through Priment that has been assessed to ensure that adequate processes are in place and are being followed for quality management, software development and security. There will be a process in place to ensure compliance and agreement with clinical trial regulations and data protection laws.

At the end of the trial the data belongs to UCL.

ELIGIBILITY:
9.1.1 TRIAL PARTICIPANT INCLUSION CRITERIA

Site Inclusion:

* FCPs must be in regular supervision
* HCPC registered Physiotherapists
* NHS patients
* Able to send monthly data uploads

Patient inclusion criteria:

* Over 18 years of age
* Registered with an included GP practice
* Consented to routine MSK data collection

9.1.2 TRIAL PARTICIPANT EXCLUSION CRITERIA

Site exclusion

* No supervision practice for FCPs
* Community service physiotherapy
* Unable to send data on a monthly basis

Patient Exclusion criteria:

* Inappropriate for FCP due to age
* Non-MSK problem
* Already managed by GP
* Unable to consent for reasons of mental health, dementia or language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Number of Participants recruited to the study | 0, 3 and 6 months
  The investigators are measuring recruitment so that we can understand the probability that we could recruit to a future trial.
Feasibility - Number of Participants retained to the study at 3 and 6 months | 3 and 6 months
  The investigators are measuring retention as a measure of retaining participants to a future trial.
Feasibility - Number of clinician participants collecting data through a template. | 3 and 6 months
  The investigators are measuring engagement with a template to assess the feasibility of participants collecting data this way in a future trial. We will report the proportion of patients whose data was collected through a template.
Feasibility of participants engaging with the dashboard intervention in a future trial | 3 and 6 months
  The investigators are measuring engagement with the dashboard through collecting logins and pages visted and time spent on the dashboard for each user, as a measure of feasibility of a future trial.
Feasibility of recording the number of clinical supervision sessions that utilise the PRISM dashboard as recorded in a supervision log | 3 and 6 months
  The investigators are measuring use of the intervention in clinical supervision via a supervision log, as a measure of feasibility of a future trial.
Completion of outcomes as a measure of feasibility | 0,3 and 6 months
  The feasibility of collecting outcomes at each time point and the rate of completion of outcomes will give the investigators a measure of how feasible it will be to collect outcomes at a future trial. A completion rate for each outcome will be reported.

SECONDARY OUTCOMES:
Clinical Decision making data points | 3 and 6 months.
  We will report proportions for each data point for groups and individual clinicians
Clinical Supervision Log | 3 and 6 months.
  We will report adherence to structured clinical supervision as a binary. Structured supervision is described in the intervention as supervision that engages with the PRISM dashboard as a learning tool.
Manchester scale of supervision | 0 3 and 6 months
  PROM on clinician experience of supervision. he MCSS-26 is a 26-item questionnaire developed specifically for clinical supervision research and evaluation. A higher score indicates a more positive experience.
EQ5D5L | 0,3 and 6 months
  The EuroQol 5-Dimension 5-Level scale. It is a standardised instrument used to measure health-related quality of life (HRQoL), widely applied in clinical trials, population health surveys, and economic evaluations of healthcare. Scoring is from 0 to 100, Higher scores indicate better health outcomes.
MSK HQ | 0,3 and 6 months
  PROM for future trial: Musculoskeletal Health Questionnaire scores from 0-56. A higher score is better MSK Health

IPD SHARING:
Plan to Share IPD: No
The data that we are processing for the trial is anonymous.

REFERENCES:
- [Background] Gould IM, Lawes T. Antibiotic stewardship: prescribing social norms. Lancet. 2016 Apr 23;387(10029):1699-701. doi: 10.1016/S0140-6736(16)00007-6. Epub 2016 Feb 18. No abstract available. PMID 26898851
- [Background] Hallsworth M, Chadborn T, Sallis A, Sanders M, Berry D, Greaves F, Clements L, Davies SC. Provision of social norm feedback to high prescribers of antibiotics in general practice: a pragmatic national randomised controlled trial. Lancet. 2016 Apr 23;387(10029):1743-52. doi: 10.1016/S0140-6736(16)00215-4. Epub 2016 Feb 18. PMID 26898856
- [Background] Tang MY, Rhodes S, Powell R, McGowan L, Howarth E, Brown B, Cotterill S. How effective are social norms interventions in changing the clinical behaviours of healthcare workers? A systematic review and meta-analysis. Implement Sci. 2021 Jan 7;16(1):8. doi: 10.1186/s13012-020-01072-1. PMID 33413437
- [Background] Ivers N, Jamtvedt G, Flottorp S, Young JM, Odgaard-Jensen J, French SD, O'Brien MA, Johansen M, Grimshaw J, Oxman AD. Audit and feedback: effects on professional practice and healthcare outcomes. Cochrane Database Syst Rev. 2012 Jun 13;2012(6):CD000259. doi: 10.1002/14651858.CD000259.pub3. PMID 22696318
- [Background] Gagliardi AR, Wright FC. Exploratory evaluation of surgical skills mentorship program design and outcomes. J Contin Educ Health Prof. 2010 Winter;30(1):51-6. doi: 10.1002/chp.20056. PMID 20222034
- [Background] Brink P, Back-Pettersson S, Sernert N. Group supervision as a means of developing professional competence within pre-hospital care. Int Emerg Nurs. 2012 Apr;20(2):76-82. doi: 10.1016/j.ienj.2011.04.001. Epub 2011 May 28. PMID 22483002
- [Background] Langridge N. The skills, knowledge and attributes needed as a first-contact physiotherapist in musculoskeletal healthcare. Musculoskeletal Care. 2019 Jun;17(2):253-260. doi: 10.1002/msc.1401. Epub 2019 Apr 17. PMID 30993860
- [Background] Physiotherapists CSo. Principles of first contact physiotherapy: a resource to support service evaluation. 2021.
- [Background] England N. Multi-professional framework for advanced clinical practice in England. 2017.
- [Background] Stynes S, Jordan KP, Hill JC, Wynne-Jones G, Cottrell E, Foster NE, Goodwin R, Bishop A. Evaluation of the First Contact Physiotherapy (FCP) model of primary care: patient characteristics and outcomes. Physiotherapy. 2021 Dec;113:199-208. doi: 10.1016/j.physio.2021.08.002. Epub 2021 Aug 6. PMID 34656297
- [Background] Goodwin R, Moffatt F, Hendrick P, Stynes S, Bishop A, Logan P. Evaluation of the First Contact Physiotherapy (FCP) model of primary care: a qualitative insight. Physiotherapy. 2021 Dec;113:209-216. doi: 10.1016/j.physio.2021.08.003. Epub 2021 Aug 6. PMID 34583834
- [Background] England N. The NHS Long Term Plan 2019.
- [Background] UK D. The Musculoskeletal Services Framework-A joint responsibility: doing it differently. Health, Editor. 2006:72.
- [Background] Keavy R. The prevalence of musculoskeletal presentations in general practice: an epidemiological study. Br J Gen Pract. 2020 Jun;70(suppl 1):bjgp20X711497. doi: 10.3399/bjgp20X711497. PMID 32554673